CLINICAL TRIAL: NCT03769285
Title: Nicotinamide Chemoprevention for Keratinocyte Carcinoma in Solid Organ Transplant Recipients: A Pilot, Placebo-controlled, Randomized Trial
Brief Title: Skin Cancer Prevention With Nicotinamide in Transplant Recipients - Pilot Trial
Acronym: SPRINTR-Pilot
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Kidney Foundation of Canada (Other); NOW Foods (Other); Natural Life Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPRINTR-Pilot
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Non-melanoma Skin Cancer; Carcinoma, Squamous Cell; Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Nicotinamide — Oral nicotinamide (500 mg) twice daily for at least 52 weeks
  Other Names: niacinamide
  Arms: Nicotinamide
Drug: Placebo oral capsule — Matching placebo taken twice daily for at least 52 weeks
  Arms: Placebo

SUMMARY:
A common long-term side effect of anti-rejection (immunosuppressant) medications is skin cancer. This pilot clinical trial evaluates the feasibility of conducting a larger pivotal trial to examine the efficacy and safety of nicotinamide for prevention of keratinocyte carcinoma in solid organ transplant recipients. This pilot trial will transition into the pivotal trial if all feasibility targets are met.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Kidney, liver, heart, or lung transplant at least two years ago
3. History of at least one prior histologically-confirmed keratinocyte carcinoma or squamous cell carcinoma in situ
4. Currently immunosuppressed with a calcineurin inhibitor-based regimen (cyclosporine or tacrolimus)
5. Able to attend follow-up visits
6. Able to speak and understand English (only for cognitive substudy)

Exclusion Criteria:

1. Use of mTOR inhibitor (sirolimus, everolimus) within the past 12 weeks
2. Biopsy-confirmed acute rejection episode within the past 12 weeks
3. Active liver disease (elevated AST or ALT >3 times normal)
4. Severe renal failure (estimated glomerular filtration rate <20 mL/min/1.73 m2)
5. Current carbamazepine or primidone use
6. Pregnancy and lactation
7. Gorlin syndrome or other genetic skin cancer syndrome
8. Solid organ or hematologic malignancy, invasive Stage II melanoma, Merkel cell carcinoma, or metastatic skin cancer within the past five years, or invasive Stage I melanoma within the past two years
9. Untreated localized skin cancer (invasive squamous cell carcinoma, basal cell carcinoma, or keratoacanthoma) at baseline (the patient can enrol after skin cancer treatment)
10. Use of nicotinamide or niacin (250 mg or more daily) within the past 12 weeks
11. Use of field therapy for actinic keratoses within the past 12 weeks
12. Initiation of systemic chemoprevention within the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility (pertaining to patient recruitment) | 1 year
  Proportion of patients who consent to data linkage to provincial administrative databases
Feasibility (pertaining to appropriateness of eligibility criteria) | 1 year
  Reasons for exclusion of screened patients
Feasibility (pertaining to adherence to intervention) | 1 year
  Proportion of capsules returned, reasons for non-adherence
Feasibility (pertaining to adherence to follow-up assessments) | 1 year
  Proportion of missed assessments and incomplete questionnaire data variables, proportion of patients who withdraw from the trial, patient perception of trial participation
Feasibility (pertaining to data linkage) | 1 year
  Proportion of patients who consent to data linkage to provincial administrative databases
Preliminary pooled keratinocyte carcinoma event rate | 1 year
  Pooled keratinocyte carcinoma event rate to be used for sample size re-estimation in the pivotal trial.
Drug interactions | 1 week
  Proportion of patients with a clinically relevant increase in cyclosporine or tacrolimus blood concentration at 1 week. An increased level will be classified as clinically relevant if the transplant physician reduces the immunosuppressant dose in response to the increased drug level.
Drug interactions | 2 weeks
  Proportion of patients with a clinically relevant increase in cyclosporine or tacrolimus blood concentration at 2 weeks. This measurement will be dropped if all cases of clinically relevant drug interactions manifest at 1 week in the first 20 enrolled participants.
Serious adverse events | 1 year
  Descriptive tabulation (preliminary safety)

SECONDARY OUTCOMES:
Feasibility of recruiting for neurocognitive substudy | 1 year
  Proportion of enrolled participants who consent to participate in the neurocognitive substudy
Baseline prevalence of cognitive impairment (substudy) | 1 year
  Montreal Cognitive Assessment (MoCA) score <26, scored out of 30.
Pooled standard deviation of MoCA test scores (substudy) | 1 year
  Montreal Cognitive Assessment (MoCA), raw scores are scored out of 30, with a higher score representing better cognitive function
Pooled standard deviation of Hopkins Verbal Learning Test - Revised scores (substudy) | 1 year
  Hopkins Verbal Learning Test - Revised, a memory test scored out of 60, with a higher score representing better memory
Pooled standard deviation of Trail Making A and B test scores (substudy) | 1 year
  Trail Making A and B, a visual attention test. This records the time (in seconds) to completion, with a faster time representing better cognitive function
Pooled standard deviation of Controlled Oral Word Association test scores (substudy) | 1 year
  Controlled Oral Word Association, a verbal fluency test, measures the production of words belonging to the same letter. This records total number of words produced, with a higher number representing better verbal fluency.
Pooled standard deviation of Animal Naming Task scores (substudy) | 1 year
  Animal Naming Task, a verbal fluency task, measures the total number of animals named in one minute, with a higher number representing better verbal fluency
Pooled standard deviation of cognitive test scores (substudy) | 1 year
  Wechsler Adult Intelligence Scale - Revised, Digit Span subtest, a number sequencing memory test, measures the number of correctly repeated sequences with maximum score of 48. The higher score represents better cognitive function
Pooled standard deviation of serum phosphate levels (substudy) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: An-Wen Chan, MD DPhil, Principal Investigator — Women's College Hospital; Joseph Kim, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
If feasibility thresholds are met, this pilot trial will proceed to a larger pivotal trial. The study protocol for the pivotal trial will be published prior to completion of data collection. Beyond 2 years after completion of the pivotal trial, the cleaned, anonymized, participant-level dataset and statistical code will made available for sharing with external researchers upon approval of a study proposal describing the intended data usage.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2 years after completion of the pivotal trial that follows this pilot trial